CLINICAL TRIAL: NCT06655220
Title: Investigation of the Effect of BI 1815368 on the Pharmacokinetics of Metformin Following Multiple Oral Administration in Healthy Subjects (an Open-label, Randomised, Two-way Crossover Trial)
Brief Title: A Study in Healthy Men to Test Whether BI 1815368 Influences the Amount of Metformin in the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1485-0013; 2024-515911-23-00 (Other: CTIS); U1111-1306-9403 (Other: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Two-way crossover trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin hydrochloride alone (reference) followed by metformin hydrochloride + BI 1815368 (Test) (Experimental)
  Interventions: Drug: Metformin hydrochloride; Drug: BI 1815368
- Metformin hydrochloride + BI 1815368 (Test) followed by metformin hydrochloride alone (reference) (Experimental)
  Interventions: Drug: Metformin hydrochloride; Drug: BI 1815368

INTERVENTIONS:
Drug: Metformin hydrochloride — Metformin hydrochloride
Drug: BI 1815368 — BI 1815368

SUMMARY:
The main objective of this trial is to investigate the effect on the exposure of metformin in plasma when administered as an oral multiple dose together with multiple oral doses of BI 1815368 (Test, T) as compared to when metformin is administered as an oral multiple dose alone (Reference, R).

ELIGIBILITY:
Inclusion criteria:

1. Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
2. Age of 18 to 50 years (inclusive)
3. Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
4. Signed and dated written informed consent in accordance with international conference on harmonization-good clinical practice (ICH-GCP) and local legislation prior to admission to the trial

Exclusion criteria:

1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
6. Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
7. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
8. History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2024-11-08 (Actual); Primary Completion 2024-12-08 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
AUC τ,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ) | Up to 2 days after last dose administration
C max,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | Up to 2 days after last dose administration

SECONDARY OUTCOMES:
CL R,ss (renal clearance of the analyte from plasma at steady state) | Up to 2 days after last dose administration

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com